CLINICAL TRIAL: NCT03426254
Title: Comparison of Safety and Clinical Benefit of Injections Subcutaneously Talazoparib Versus Oral Talazoparib in Patients With Advanced Solid Tumors ( Phase I )
Brief Title: Comparison of Safety and Clinical Benefit of Injections Subcutaneously Talazoparib Versus Oral Talazoparib in Patients With Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: the company is liquidated
Sponsor: Center Trials & Treatment (Other)
Collaborators: BioGene Pharmaceutical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TST-9-H
Record Dates: First submitted 2018-01-27; First posted 2018-02-08 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Advanced or Recurrent Solid Tumors; Breast Neoplasm
Keywords: Subcutaneously Talazoparib
MeSH Terms: conditions — Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Intervention Model Description: The intent of this study was to assess the safety and efficacy of two forms of Talazoparib therapy for the treatment of advanced solid tumors . After an enrollment period, patients will randomized to receive oral Talazoparib (1 mg, one times a day ) or subcutaneously Talazoparib (1 mg subcutaneous injection by pen-syringe / mechanical dispenser) .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injections Subcutaneously Talazoparib (Experimental): Patients receive per day single dose of subcutaneous Injection contains 1 mg Talazoparib on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Auto-Injector delivers a single dose of 1 mg Talazoparib injection (subcutaneous)
  Interventions: Biological: Injections Subcutaneously Talazoparib
- Oral capsules Talazoparib (Active Comparator): Patients receive 1 mg of Talazoparib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Oral capsules Talazoparib

INTERVENTIONS:
Biological: Injections Subcutaneously Talazoparib — Patients receive per day single dose of subcutaneous Injection contains 1 mg Talazoparib on days 1-28
  Other Names: MDV3800; BMN673
  Arms: Injections Subcutaneously Talazoparib
Drug: Oral capsules Talazoparib — Patients receive 1 mg of Talazoparib PO QD on days 1-28.
  Other Names: MDV3800; BMN673
  Arms: Oral capsules Talazoparib

SUMMARY:
To assess the safety and efficacy of two forms of Talazoparib therapy (injections subcutaneously Talazoparib and oral form for the treatment in the equivalent therapeutics dose

DETAILED DESCRIPTION:
The intent of this study was to assess the safety and efficacy of two forms of Talazoparib therapy for the treatment of advanced solid tumors . After an enrollment period, patients will randomized to receive oral Talazoparib (1 mg, one times a day ) or subcutaneously Talazoparib (1 mg by subcutaneous injection with NovoPen / Autopen) one times a day in the appropriate volume

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form (by the patient or a legally acceptable representative as per the local regulations) obtained prior to initiation of any study-specific procedure and treatment.
* Female of at least 21 years of age.
* Histologically or cytologically confirmed advanced solid tumor with no available standard approved treatment options in the opinion of the Investigator
* Eastern Cooperative Oncology Group (ECOG) Performance status (PS) ≤ 2.
* Renal function at screening and enrollment as defined by the
* Patient has had no clinically significant change in renal status within 3 months prior to screening, according to Investigator's review of clinical patient records.
* Patient is not currently on hemodialysis and/or peritoneal dialysis for management of chronic kidney disease or acute failure/conditions.
* Patient has no unstable renal function, defined as a change in estimated glomerular filtration rate (eGFR) (calculated with the MDRD equation) of > 25% for patients with mild and moderate renal impaired or as a change in eGFR > 30% for patients with severe renal impaired, from screening to enrollment.
* Received at least 1 and no more than 3 platinum-based chemotherapy regimens (prior bevacizumab is allowed) and the last dose is ≥ 28 days before randomization
* No prior PARP inhibitor treatment
* Adequate other organ function at screening and enrollment.
* Female patients of childbearing potential must have a negative serum pregnancy test at screening, and must agree to use a highly effective birth control method from the time of the first dose of study drug through 60 days after the last dose of study drug.
* Female patients must not be breastfeeding at screening nor during the study participation until 60 days after the last dose of study drug.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Terminology Criteria for Adverse Events [CTCAE] grade ≤ 1) from the acute toxicities of previous therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting eligibility requirements.
* Use of any investigational agent within 14 days before randomization.
* Had > 2 paracentesis procedures within 28 days before randomization.
* Major surgery within 14 days before randomization.
* Requirement for intravenous alimentation (at the time of randomization).
* Seropositive for human immunodeficiency virus (HIV).
* Any serious or unstable medical condition that interferes with ability to tolerate treatment or assessments associated with the protocol.
* Gastrointestinal disorder affecting absorption.
* Known or suspected hypersensitivity to any of the talazoparib capsule components.
* Any condition or reason that interferes with ability to participate in the study, tolerate treatment or assessments associated with the protocol, causes undue risk, or complicates the interpretation of safety data, in the opinion of the Investigator or Medical Monitor.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-10 (Estimated); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of occurrence and evaluation of adverse events in the use of Subcutaneously Talazoparib ( 1 mg / dose ) | Anticipated in about 12 month following first patient enrolled
  Frequency of occurrence and evaluation of adverse events in the use of Subcutaneously Talazoparib , assessed by percentage of patients with any Adverse Event (AE), leading to Study Drug Discontinuation, Serious Adverse Event (SAE), related to study drug, SAE related to study drug.
  Incidence of toxicity, graded according to the National Cancer Institute (NCI) CTCAE version 4.03 Incidence of toxicity, graded according to the National Cancer Institute (NCI) CTCAE version 4.03

SECONDARY OUTCOMES:
Clinical Benefit of Injections Subcutaneously Talazoparib | Every 9 weeks for 12 months
  Clinical benefit (CB) defined as any of the following, complete response, partial response, or stable disease for > 24 weeks by RECIST 1.1. Assessments performed using computed tomography (CT) or magnetic resonance imaging (MRI) or ultrasound examination (Use) scan every 9 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- University -Mother Theresa- Hospital, Oncology Dep., Tirana, Albania